CLINICAL TRIAL: NCT00559611
Title: Prospective Comparison of Endobronchial Ultrasound Needle Biopsy Versus Mediastinoscopy for Staging of Mediastinal Nodes in Patients With Clinical Stage IIIA Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Endobronchial Ultrasound Versus Mediastinoscopy in Patients With Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-0353; NCI-2011-01302 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Lung Cancer
Keywords: Non-Small Lung Cancer; Lung Cancer; Endobronchial Ultrasound; Fine Needle Aspiration; Mediastinoscopy; EBUS-FNA; EBUS; Needle Biopsy; NSCLC
MeSH Terms: conditions — Lung Neoplasms | interventions — Mediastinoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- Endobronchial Ultrasound vs. Mediastinoscopy (Experimental): Endobronchial Ultrasound - A small flexible scope is passed down the windpipe. Samples of lymph gland tissue will be collected through a tiny needle that is passed through the scope.
  Mediastinoscopy - Performed if a tumor is not found on the opposite side of your chest from another tumor by the EBUS.
  Interventions: Procedure: Endobronchial Ultrasound; Procedure: Mediastinoscopy

INTERVENTIONS:
Procedure: Endobronchial Ultrasound — A small flexible scope is passed down the windpipe. Samples of lymph gland tissue will be collected through a tiny needle that is passed through the scope.
  Other Names: EBUS
Procedure: Mediastinoscopy — Performed if a tumor is not found on the opposite side of your chest from another tumor by the EBUS.

SUMMARY:
The goal of this clinical research study is to compare 2 different methods for checking lymph glands (in the middle of the chest) for cancer cells.

Objectives:

The aim of this prospective study is to determine the staging accuracy of endobronchial ultrasound guided fine needle aspiration biopsy of mediastinal lymph nodes compared to the 'gold standard', mediastinoscopy, in patients with clinical Stage IIIA non-small cell lung cancer.

Primary Objective:

To determine the sensitivity, specificity, positive predictive value, negative predictive value, and accuracy of EBUS-FNA and mediastinoscopy in identifying mediastinal nodal metastases.

Secondary Objectives:

To estimate quantitative and qualitative differences regarding sampling of mediastinal nodes (number and location of nodes biopsied, number and location of positive nodes, extracapsular extension, ability to biopsy contralateral nodes).

To determine the frequency of change of planned therapeutic management resulting from outcome of EBUS-FNA and mediastinoscopy.

To determine procedure related complications. To perform analysis of cost between EBUS-FNA and mediastinoscopy.

DETAILED DESCRIPTION:
The current procedure used to check for cancer cells in the lungs is a small operation at the base of the neck (mediastinoscopy) to get samples of the lymph glands. These samples are then looked at under the microscope to see if they contain cancer cells. A procedure has been developed that may allow doctors to get samples of lymph glands without having to perform an operation. This is called endobronchial ultrasound or "EBUS". The purpose of this study is to compare the 2 procedures.

If you agree to take part in this study, your insurance provider will be contacted. In order for you to take part in this study, your insurance provider must agree to pay for both the EBUS and mediastinoscopy procedures.

If your insurance provider agrees to pay for both procedures, you will be scheduled for the EBUS and a mediastinoscopy. The procedures will not be scheduled on the same day. You will first have the EBUS. You will receive general anesthesia and a small flexible scope will be passed down your windpipe. Samples of your lymph gland tissue will then be collected through a tiny needle that is passed through the scope. This will be performed as an out patient procedure.

If a tumor is found on the opposite side of your chest from another tumor by the EBUS, a mediastinoscopy will not be necessary.

If a tumor is not found on the opposite side of your chest from another tumor by the EBUS, you will then have a mediastinoscopy. This is also an outpatient procedure that will involve a small (2 cm) cut at the base of the neck, just above the breast bone. Your doctor will then pass a special scope with a camera into your chest (below the breast bone). This will allow your doctor to see the lymph glands around your windpipe and get samples of them. This will also be performed under general anesthesia and you will be able to leave the hospital shortly after the procedure.

Depending on whether or not the lymph glands have cancer in them, your doctor will then recommend the best therapy for the tumor to you.

This is an investigational study. The EBUS is FDA approved. The mediastinoscopy is considered standard of care. The comparison of the 2 procedures is investigational.

Up to 100 patients will be take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be >/= 18 years old.
2. Patient must have ECOG/Zubrod status 0, 1, or 2.
3. Patient must have clinically resectable, NSCLC (squamous cell, adenocarcinoma, sarcomatoid, neuroendocrine or large cell) and be clinical Stage IIIa, according to the 1998 staging system of the American Joint Commission on Cancer for lung cancer.
4. Patient must have proven or suspected NSCLC prior to registration. Patients who obtain subsequent pathologic confirmation of NSCLC at the time of EBUS or subsequent surgery will remain enrolled on the study. Patients subsequently found to have an etiology other than NSCLC will be excluded from further analysis.
5. Patient must be anticipated to have definitive therapy for primary NSCLC. This may include surgery, chemotherapy, radiation therapy or a combination the above.
6. Patient must be medically fit for definitive therapy.
7. Patient or the patient's legally acceptable representative must provide a signed and dated written informed consent prior to registration and any study-related procedures.

Exclusion Criteria:

1. Patient has received prior chemotherapy or radiotherapy for this cancer.
2. Patient is considered a poor risk due to non-malignant systemic disease (cardiovascular, renal, etc.) that would preclude the treatment options.
3. Patient has contraindication to either endobronchial ultrasound or mediastinoscopy such as: Latex allergy; Bleeding diathesis; Previous mediastinoscopy; Previous mediastinal nodal resection; Previous tracheostomy.
4. Patients malignancy not consistent with NSCLC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2007-10-19 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
Number Patients Restaged Upwards by Mediastinoscopy Following EBUS Evaluation | 2 Years
  Outcome defined as how many patients EBUS stage N0/1 actually end up being N2/3, and how many EBUS stage N2 actually are N3 by mediastinoscopy. Study primarily interested in an upper limit on this proportion. Primary analysis is the upper one-sided 90% confidence limit.

CONTACTS AND LOCATIONS:
Overall Officials: David C. Rice, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org